CLINICAL TRIAL: NCT01628302
Title: Investigation of Salt Restriction Effect on Renin Activation
Brief Title: Effect of Salt Restriction on Renin Activation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turkish Society of Hypertension and Renal Diseases (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HT-Salt
Record Dates: First submitted 2012-06-13; First posted 2012-06-26 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2011-08

CONDITIONS: Hypertension
Keywords: Hypertension,plasma renin activity,salt consumption
MeSH Terms: conditions — Hypertension | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal salt diet (No Intervention): The group had normal salt diet (250mmol)for three weeks. Subjects had normal salt diet in their daily routine life for the following 2 weeks.According to crossover nature of the study, the group had low salt diet (50mmol) at the last 3 weeks of the study.
- Low salt diet (Experimental): The group had low salt diet (50mmol)for three weeks. Subjects had normal salt diet in their daily routine life for the following 2 weeks.According to crossover nature of the study, the group had normal salt diet at the last 3 weeks of the study.
  Interventions: Behavioral: Lowering salt in diet

INTERVENTIONS:
Behavioral: Lowering salt in diet — Low salt diet (50mmol)for three weeks.
  Arms: Low salt diet

SUMMARY:
The present prospective, randomized, crossover study is designed to investigate the effect of salt consumption on blood pressure in hypertensive subjects.

Secondary objectives of the study are to evaluate the effect of salt consumption on blood pressure among the subjects who are hypertensive and obese and normal according to body mass index and to evaluate the effect of salt consumption on renin activity in hypertensive subjects.

DETAILED DESCRIPTION:
The present study is carried out with the subjects who are chosen among the nursing home residents in İzmir. The subjects were randomized to 2 groups and while one of these groups had low salt diet (50mmol), the other group had normal salt diet (250mmol) for 3 weeks. Subjects had normal salt diet in their daily routine life for the following 2 weeks. According to crossover nature of the study, the group that had normal salt diet at the first 3 weeks of study had low salt diet at the last 3 weeks of the study. The other group that had low salt diet had the normal salt diet at the last 3 week of the study.

At the beginning of the study, information such as demographic, family story, medical story, diet habits, concomitant medication and physical measurements (height, weight and waist circumference) were received from the subjects.

24 hour blood pressure of the subjects is measured for four times, before the beginning of diet specific to their groups, at the end of the 3-week diet, before the beginning of the second diet and at the end of their second diet. The subjects were asked for collecting 24-h urine in the same days of blood pressure measurement. Sodium, potassium, urea, creatinin and microalbumin measurements were measured in the collected urine. Blood samples were collected for three times, at the end of the 3-week diet, before the beginning of the second diet and at the end of their second diet. Plasma renin activity and aldosterone levels were measured in the blood samples collected. Aldosterone level was measured in the 24-hour urine in mentioned days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are 50 years and older
* Subjects whose systolic blood pressure is ≥ 140 mmHg
* Subjects whose diastolic blood pressure is ≥ 90 mmHg
* Subjects who is normal weighted defined as body mass index < 25 or who is obese defined as body mass index > 30
* Subjects who have intellectual capacity to adapt diets and 24 hour urine collection
* Informed about the study and consented to include the study

Exclusion Criteria:

* Known heart failure
* Known renal failure
* Known chronic liver disease
* Antihypertensive drug use
* nonsteroidal anti inflammatory (NSAI) drug use

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in 24-hour ambulatory blood pressure at 3 weeks | 3 weeks
  24-hour ambulatory blood pressure was measured before the beginning of diet specific to their groups, at the end of the 3-week diet, before the beginning of the second diet and at the end of their second diet.

SECONDARY OUTCOMES:
Change in sodium levels in urine samples. | 3 weeks
  Sodium was measured in 24-hour collected urine samples before the beginning of diet specific to their groups, at the end of the 3-week diet, before the beginning of the second diet and at the end of their second diet.
Change in plasma renin activity | For 3 times in 8 weeks
  Plasma renin activity level was measured in the blood samples collected, at the end of the 3-week diet, before the beginning of the second diet and at the end of their second diet.
Change in aldosterone level in blood samples | For 3 times in 8 weeks
  Aldosterone levels was measured in the blood samples collected , at the end of the 3-week diet, before the beginning of the second diet and at the end of their second diet.
Change in potassium levels in urine samples. | 3 weeks
  Potassium was measured in 24-hour collected urine samples before the beginning of diet specific to their groups, at the end of the 3-week diet, before the beginning of the second diet and at the end of their second diet.
Change in urea level in urine samples | 3 weeks
  Urea was measured in 24-hour collected urine samples before the beginning of diet specific to their groups, at the end of the 3-week diet, before the beginning of the second diet and at the end of their second diet
Change in creatinin level in urine samples | 3 weeks
  Creatinin was measured in 24-hour collected urine samples before the beginning of diet specific to their groups, at the end of the 3-week diet, before the beginning of the second diet and at the end of their second diet.
Change in microalbumin level in urine samples | 3 weeks
  Microalbumin was measured in 24-hour collected urine samples before the beginning of diet specific to their groups, at the end of the 3-week diet, before the beginning of the second diet and at the end of their second diet
Change in aldosterone level in urine samples | For 3 times in 8 weeks
  Aldosterone levels was measured in in the 24-hour urine samples collected , at the end of the 3-week diet, before the beginning of the second diet and at the end of their second diet.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Arici, Prof., Principal Investigator — Hacettepe University Faculty of Medicine Department of Nephrology